CLINICAL TRIAL: NCT03333655
Title: A Multicenter Study to Explore the Mechanism of Acquired Immune Escape In Patients With Metastatic Cancer Progressing on Checkpoint Inhibitor Therapy
Brief Title: Study to Explore the Mechanism of Acquired Immune Escape In Participants With Metastatic Cancer Progressing on CPI Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ML40108
Record Dates: First submitted 2017-10-04; First posted 2017-11-07 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Neoplasms
Keywords: Metastatic Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Checkpoint Inhibitor Therapy (Other): Pre-treatment (archival) and at progression biopsy for participants with a demonstrated clinical benefit on CPI therapy will be asked to participate in the study. In addition, retrospective enrollment of patients who progressed on CPI therapy after documented response and for whom an at-progression biopsy is available, is also possible.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Participants who received or are receiving CPI therapy for metastatic cancer or hematologic malignancies.

SUMMARY:
The purpose of this study is to identify mechanisms associated with acquired immune escape by comparing baseline and at-progression tissue samples from participants who derive clinical benefit from CPI treatment of metastatic cancer or hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Response assessment of complete response (CR), partial response (PR), or long-term stable disease (SD) for >6 months with a cancer immunotherapy treatment for metastatic cancer or hematologic malignancies either through a marketed CPI or through participation in a Roche/Genentech CPI clinical trial.
* Availability of tissue sample.

Exclusion Criteria:

* Pregnant, lactating, or intending to become pregnant during the study.
* Participants receiving CPI treatment as part of a non-Roche/Genentech clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Number of Gene Alterations in at-Progression Biopsy of Patricipants with Acquired Immune Escape | Day 1
  Number of Gene Alterations Will Be Evaluated Using NGS Approaches by Comparing At-Progression Biopsy with Pre-Treatment Biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (11):
- United States (5):
  - UCSF Comp Canc Ctr, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine; Dept of Medicine/Div of Medical Oncology, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center; Herbert Irving Pavillion, New York, New York
  - Sarah Cannon Cancer Center, Arrington, Tennessee
- Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse, France
- South Korea (2):
  - Seoul National University Hospital; Department of Oncology, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
- Spain (2):
  - Clinica Universitaria de Navarra; Servicio de oncología, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
- Barts Hospital; Institute of Cancer, London, United Kingdom